CLINICAL TRIAL: NCT05224648
Title: Comparison of Train of Four, Tetanus 50 Hz and Tetanus 100 Hz Recovery Following Rocuronium Induced Neuromuscular Block Reversed by Neostigmine
Brief Title: Comparison of Train of Four, Tetanus 50 and 100 Hz Recovery After Rocuronium Block Reversed by Neostigmine
Acronym: DECURATOF 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DECURATOF 2
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Residual Curarization
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOF scan train of four ratio monitoring (Active Comparator): recovery of train of four ratio after neostigmine administration
  Interventions: Device: TOF scan train of four ratio monitoring
- ITF device tetanus stimulation monitoring (Experimental): recovery of tetanus 100 Hz and tetanus 50 Hz ratio after neostigmine administration
  Interventions: Device: ITF device tetanus stimulation monitoring

INTERVENTIONS:
Device: TOF scan train of four ratio monitoring — Device : TOF Scan For each included patient, 2 monitorings (TOF Scan and ITF device) will be placed, one on each hand. Once 4 contractions of the adductor pollicis muscle will be observed on the TOF Scan side following train of four stimulation, 40 µg/kg neostigmine will be injected. Train of four ratio (delivered every minute) will be recorded. This sequence (tetanus 100 Hz followed by tetanus 50 Hz) will be repeated 6 times. For each tetanus stimulation, the ratio between the residual force and the maximum force generated by the adductor pollicis muscle will be recorded (this ratio illustrates the fade phenomenon). At the end of this period lasting 30 minutes after neostigmine administration, anesthetic drug delivery will be stopped and the patient wil be allowed to recover.
  Arms: TOF scan train of four ratio monitoring
Device: ITF device tetanus stimulation monitoring — Device ITF For each included patient, 2 monitorings (TOF Scan and ITF device) will be placed, one on each hand. Once 4 contractions of the adductor pollicis muscle will be observed on the TOF Scan side following train of four stimulation, 40 µg/kg neostigmine will be injected. Train of four ratio (delivered every minute) will be recorded. This sequence (tetanus 100 Hz followed by tetanus 50 Hz) will be repeated 6 times. For each tetanus stimulation, the ratio between the residual force and the maximum force generated by the adductor pollicis muscle will be recorded (this ratio illustrates the fade phenomenon). At the end of this period lasting 30 minutes after neostigmine administration, anesthetic drug delivery will be stopped and the patient wil be allowed to recover.
  Arms: ITF device tetanus stimulation monitoring

SUMMARY:
Despite neuromuscular transmission monitoring and pharmacological reversal allowing a train of four ratio recovery higher than 0.9, patients receiving neuromuscular blocking agent during general anesthesia have a high risk of postoperative pulmonary complications. While this train of four ratio threshold is considered as the gold standard to confirm the lack of residual paralysis, tetanus 100 Hz stimulation showed a marked fade. This result has been observed in absence of reversal agent administration.

Therefore, the present study has been designed to compare the recovery of train of four stimulation, tetanus 50 Hz and tetanus 100 Hz stimulation in patient receiving rocuronium during general anesthesia and reversed by an anticholinesterase agent (neostigmine). Neostigmine will be injected once four muscular contractions of the adductor pollicis muscle will be observed after a train of four stimulation, at a dose (40 µg/kg) in accordance with the clinical practice worldwide admitted.

Two questions have to be investigated. First, is this dose of neostigmine sufficient to allow a complete recovery of tetanus stimulations ? Second, due to the pharmacological properties of neostigmine, does a recurarisation phenomenon occur following repeated tetanus stimulations ? The attented results of this study will be to propose a new thinking on what we really need to make relevant progress in the safety aspects of residual paralysis outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA clinical status 1 to 3 informed consent obtained before anesthesia induction

Exclusion Criteria:

* ASA clinical status 4 emergency surgery scheduled surgery in prone position hepatic or renal disease BMI higher than 35 allergy to rocuronium or neostigmine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
To determine the delay following neostigmine administration to obtain a train of four ratio higher than 0.9 and a tetanus 100 Hz ratio higher than 0.9 | 30 minutes after neostigmine administration

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Debaene, MD phD, Study Director — CHU de Poitiers FRANCE
Locations (1):
- CHU de Poitiers, Poitiers, France